CLINICAL TRIAL: NCT00986557
Title: A Randomised Controlled Phase II Trial of the Adoptive Transfer of Selected Cytomegalovirus-Specific Cytotoxic T Lymphocytes (CMV-CTL) After Allogeneic Stem Cell Transplantation (SCT) in Patients at Risk of CMV Disease
Brief Title: T-Lymphocyte Infusion or Standard Therapy in Treating Patients at Risk of Cytomegalovirus Infection After a Donor Stem Cell Transplant
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Birmingham (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000650654; CRC-TU-ACE-CMV; 53325562; EU-20974
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2010-04

CONDITIONS: Graft Versus Host Disease; Nonneoplastic Condition
Keywords: cytomegalovirus infection; graft versus host disease
MeSH Terms: conditions — Graft vs Host Disease; Cytomegalovirus Infections | interventions — Immunotherapy, Adoptive; Alemtuzumab; Foscarnet; Ganciclovir; Polymerase Chain Reaction; Therapeutics; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: adoptive immunotherapy
Biological: alemtuzumab
Biological: in vitro-treated peripheral blood lymphocyte therapy
Drug: foscarnet sodium
Drug: ganciclovir
Genetic: polymerase chain reaction
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: infection prophylaxis and management
Procedure: peripheral blood stem cell transplantation
Procedure: standard follow-up care
Radiation: radiation therapy

SUMMARY:
RATIONALE: An infusion of cytomegalovirus-specific T lymphocytes may prevent or reduce cytomegalovirus infection during the first year after a donor stem cell transplant.

PURPOSE: This randomized phase II trial is studying T-lymphocyte infusion to see how well it works compared with standard therapy in treating patients at risk of cytomegalovirus infection after a donor stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the frequency of cytomegalovirus (CMV) reactivation during the first year after allogeneic stem cell transplantation (ASCT) in patients at risk for CMV infection treated with adoptive transfer of selected CMV-specific cytotoxic T-lymphocytes.

Secondary

* To monitor CMV-specific immune reconstitution within the first year following ASCT in these patients.
* To determine the time to CMV reactivation in these patients.
* To evaluate the use of antiviral therapy in these patients.
* To determine the incidence of secondary CMV reactivation and CMV disease in patients treated with this regimen.
* To determine the incidence of acute and chronic graft-versus-host disease.

OUTLINE: This is a multicenter study. After undergoing an allogeneic peripheral blood stem cell transplantation (PBSCT) using an alemtuzumab-based conditioning regimen that also includes radiotherapy, patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive cytomegalovirus (CMV)-specific cytotoxic T-lymphocyte infusion on day 21-90 after allogeneic PBSCT.
* Arm II: Patients undergo standard follow-up care and receive standard antiviral therapy comprising ganciclovir IV or foscarnet sodium upon detection or confirmation of CMV reactivation.

Blood samples are collected to assess CMV viral load by quantitative PCR.

After completion of study therapy, patients are followed once a week for 100 days and then once a month for 1 year.

PROJECTED ACCRUAL: A total of 18 patients with sibling donors and 21 patients with unrelated donors are accrued for each arm, resulting in a total of 78 patients accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Planning allogeneic peripheral blood stem cell transplantation (PBSCT) using a conditioning regimen containing alemtuzumab and radiotherapy
* Sibling or matched unrelated donor available

  * Patients and donor matched for ≥ one of the following HLA alleles:

    * HLA-A*0101
    * HLA*0201
    * HLA-A*1101
    * HLA-A*2402
    * HLA-B*0702
    * HLA-B*0801
    * HLA-B*3502
  * No donors whose stem cells have already been collected and cryopreserved prior to transplant
* Patient and donor must be CMV seropositive
* Stem cell harvests ≥ 4.0 x 10^6 CD34 cells/kg

PATIENT CHARACTERISTICS:

* See Disease Characteristics

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior bone marrow transplantation
* No concurrent participation in another therapeutic transplantation study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2009-09; Primary Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
CMV reactivation in the first year after ASCT measured by quantitative PCR

SECONDARY OUTCOMES:
CMV-specific T-cell reconstitution by detection of circulating T-cell responses to CMV in the first year after ASCT
Time to CMV reactivation
Use of antiviral therapy
Incidence of secondary CMV reactivation and CMV disease
Incidence of acute and chronic graft-versus-host disease

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Chen, MD, Principal Investigator — University Hospital Birmingham
Locations (1):
- Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England, United Kingdom